CLINICAL TRIAL: NCT01837758
Title: Changes in Platelet Function During Continuous Veno-venous Hemodialysis Using the Multiplate Device
Brief Title: Monitoring Platelet Function During Continuous Hemodialysis
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Saskia Wand, Dr. med Saskia Wand, Goethe University
Other Study IDs: CVVH-Multiplate
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Platelet Function
Keywords: Platelet function; hemofiltration; Multiplate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dialysis: Platelet function will be documented during the first 48 hours of veno-venous hemofiltration using the Multiplate system.

SUMMARY:
Aim of the study is a description of changes in platelet function during continuous veno-venous hemodialysis or hemofiltration in patients on an intensive care unit using the Multiplate system.

ELIGIBILITY:
Inclusion Criteria:

* Need for a continuous renal replacement therapy
* Platelet Count >100.000/nl

Exclusion Criteria:

* Pregnancy
* Age <18 years
* Renal replacement therapy within the 7 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in an intensive care unit with the need for a renal replacement therapy-
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
ASPItest | Baseline, 6, 12, 24 and 48 hours
  Area under the aggregation curve (AUC) after platelet stimulation with arachidonic acid at baseline and 6, 12, 24 and 48 hours after the start of the continuous hemofiltration.

SECONDARY OUTCOMES:
ADPtest | Baseline, 6, 12, 24 and 48 hours
  Area under the aggregation curve (AUC) after platelet stimulation with adenosine diphosphate at baseline and 6, 12, 24 and 48 hours after the start of the continuous hemofiltration.
TRAPtest | Baseline, 6, 12, 24, 48 hours
  Area under the aggregation curve (AUC) after platelet stimulation with thrombin-receptor-activating peptide 6 (TRAP-6) at baseline and 6, 12, 24 and 48 hours after the start of the continuous hemofiltration.
CT-INTEM | Baseline, 6, 12, 24 and 48 hours
  Clotting time (CT) in the intrinsically activated rotational thrombelastometry (ROTEM) recorded in seconds at baseline and 6, 12, 24 and 48 hours after the start of continuous veno-venous hemofiltration.
MCF-INTEM | Baseline, 6, 12, 24 and 48hours
  Maximum clot firmness (MCF) in the intrinsically activated rotational thrombelastometry (ROTEM) recorded in millimeters at baseline and 6, 12, 24 and 48 hours after the start of continuous veno-venous hemofiltration.

OTHER OUTCOMES:
Age | Baseline
  Age of the patient at the point of enrollment
Height | Baseline
  Height of the patient measured in centimeters.
Weight | Baseline
  Weight of the patient measured in kilograms.
Gender | Baseline
ASA-Classification | Baseline
  The ASA-Classification will be determined preoperatively.
Antiaggregatory Premedication | Baseline
  Antiaggregatory medication taken prior to enrollment wil be recorded in the categories aspirin, clopidogrel, ticagrelor, cumarins and others.
Dialysis filter | Basline
  The brand of filter used for the hemofiltration or hemodialysis will be registered.
Anticoagulation for hemofiltration | Baseline
  The anticoagulation used for hemofiltration will be recorded in the categories heparin and calcium citrate.

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Daugirdas JT, Bernardo AA. Hemodialysis effect on platelet count and function and hemodialysis-associated thrombocytopenia. Kidney Int. 2012 Jul;82(2):147-57. doi: 10.1038/ki.2012.130. Epub 2012 May 16. PMID 22592187